CLINICAL TRIAL: NCT04910464
Title: Could Early Tranexamic Acid Safely Serve as an Anti-inflammatory Treatment for Patients With Sepsis? A Randomized Double Blind Controlled Trial
Brief Title: Early Tranexamic Acid and Modulating the Inflammatory Response in Sepsis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300607
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Give 1 gram of TXA in 100 ml of 0.9% normal saline, intravenous over 10 minutes as soon as possible but no later than three hours after diagnosis, infuse a second gram of TXA IV over 8 hours in 0.9% normal saline for the first 3 days.
  Interventions: Drug: Tranexamic acid
- Saline placebo (Placebo Comparator): Give the same volume (100 ml normal saline) and same duration (first three days).
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: Tranexamic acid — administer 1 gram of TXA in 100 ml of 0.9% normal saline, intravenous over 10 minutes as soon as possible but no later than three hours after diagnosis, infuse a second gram of TXA IV over 8 hours in 0.9% normal saline for first 3 days.
  Other Names: Cyclokapron
  Arms: Tranexamic acid
Other: 0.9% saline — administer the same volume (100ml normal saline) and same duration (first three days).
  Other Names: Normal saline
  Arms: Saline placebo

SUMMARY:
In this study, our aim is to investigate the role tranexamic acid in modulating inflammation in patients with sepsis.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients or their relatives.Patients will be assigned randomly to two groups (40 subjects each) with qSOFA ≥2.

In (Group T) administer 1 gram of tranexamic acid (TXA) in 100 ml of 0.9% normal saline, intravenous over 10 minutes as soon as possible but no later than three hours after diagnosis, infuse a second gram of tranexamic acid (TXA) IV over 8 hours in 0.9% normal saline for the first 3 days. In (Group C) administer the same volume (100 ml normal saline)and same duration (first three days)for controlled patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-65 years) of American society of anesthesiologists (ASA) I-II who will be diagnosed with sepsis by qSOFA ≥2
* & needed ICU admission.

Exclusion Criteria:

* Chronic renal failure
* Liver cirrhosis
* Bleeding disorders or current anticoagulant therapy
* Pregnancy or breastfeeding
* Impaired color vision
* Severe vascular ischemia, history of venous thrombosis & pulmonary embolism
* Long term treatment with acetylsalicylic acid or non-steroidal anti-inflammatory drugs not discontinued before ICU admission
* Allergy to tranexamic acid (TXA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 7days
  Short-term ICU mortality within 7days of admission and intervention

SECONDARY OUTCOMES:
Neutrophil/lymphocyte ratio (NLR) | 4 days
  From complete blood count, divide absolute number of neutrophils on lymphocyte to assess and follow up the inflammatory response in sepsis
Interleukin-6 (IL-6) serum level | 4 days
  Measurement of interleukin-6 (IL-6) serum level to assess and follow up the inflammatory response in sepsis
Glasgow coma scale (GCS) | 5 days
  Assessing the conscious level of patients by Glasgow Coma Scale (3_15)after ICU admission and intervention start give an idea on brain dysfunction in sepsis where high scores are associated with low mortality and low scores are associated with high mortality
ICU stay | 7 days
  Days of patients admission in ICU
Length of hospitalization | 7 days
  Days of patients admission in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Principal Investigator — Omar makram
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided